CLINICAL TRIAL: NCT07277218
Title: Title: Drug-coated Balloons Versus Drug-eluting Stents for the Treatment of Femoropopliteal In-Stent Restenosis: A Prospective, Multicenter, Cohort Study (The Defier Study)
Brief Title: Drug-coated Balloons Versus Drug-eluting Stents for the Treatment of Femoropopliteal In-Stent Restenosis: A Prospective, Multicenter, Cohort Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chunshui He (Other)
Collaborators: Department of Vascular Surgery, The First Affiliated Hospital of Medicine College of Zhejiang University, Hangzhou, China. (Unknown); Department of Vascular Surgery, Liyuan Hospital Affiliated Tongji Medical College of Huazhong University of Science and Technology, Wuhan, China. (Unknown); Department of Vascular Surgery, Qingdao Haici Hospital Affiliated to Qingdao University, Qingdao, China. (Unknown); Department of Vascular Surgery, School of Medicine, Affiliated Hangzhou First People's Hospital, Zhejiang University, Hangzhou, China. (Unknown); Department of Vascular Surgery, The Second Affiliated Hospital of Soochow University, Suzhou, China. (Unknown); Department of Vascular Surgery, Zhongshan Hospital, Fudan University, Shanghai, China. (Unknown); Department of Vascular Surgery, Huashan Hospital, Fudan University, Shanghai, China. (Unknown); Department of Cardiovascular Surgery, Xiamen Cardiovascular Hospital of Xiamen University, School of Medicine, Xiamen University, Xiamen, China. (Unknown); Department of Vascular Surgery, Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China. (Unknown); Biomedical Informatics and Statistics Center, School of Public Health.Fudan University, Shanghai, China. (Unknown); Department of Vascular Surgery, Xuanwu Hospital Capital MedicalUniversity, Beijing, China. (Unknown)
Responsible Party: Sponsor-Investigator, Chunshui He, Chief physician, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZY FY XGWK2
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Femoropopliteal In-Stent Restenosis (ISR)
Keywords: in-stent restenosis ; femoropopliteal artery; drug-coated balloon ; drug-eluting stent; peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug-coated Balloons vs Drug-eluting Stents for Femoropopliteal In-Stent Restenosis (Experimental)
  Interventions: Procedure: Drug-coated Balloons versus Drug-eluting Stents for the Treatment of Femoropopliteal In-Stent Restenosis

INTERVENTIONS:
Procedure: Drug-coated Balloons versus Drug-eluting Stents for the Treatment of Femoropopliteal In-Stent Restenosis — DCB Cohort: Lesions treated primarily with a paclitaxel-coated balloon, with provisional bare-metal stenting allowed for suboptimal results. DES Cohort: Lesions treated primarily with a paclitaxel-eluting stent.

SUMMARY:
Brief Summary: Defier Study What is this study about? Femoropopliteal artery disease (a type of peripheral arterial disease) often requires stenting to restore blood flow to the legs. However, a common challenge after stenting is in-stent restenosis (ISR)-the treated blood vessel narrows again over time. Two advanced treatments for ISR are available: drug-coated balloons (DCBs) and drug-eluting stents (DESs). Both deliver medication to prevent vessel narrowing, but there is limited direct evidence comparing how well they work for ISR in the femoropopliteal artery (the main artery from the thigh to the knee).

This study (called the "Defier Study") aims to fill this gap by directly comparing the safety and effectiveness of DCBs and DESs for treating femoropopliteal ISR. The results will help doctors choose the best treatment for patients with this condition.

Who can take part in the study?

Eligible patients must:

Be 18 years or older and able to provide informed consent. Have symptoms of reduced blood flow to the legs (Rutherford class 2-5, e.g., pain when walking, rest pain, or skin changes).

Have a narrowed (≥50%) or blocked femoropopliteal stent (implanted more than 30 days earlier), with the affected area no longer than 30 cm.

Have at least one open blood vessel below the knee (to ensure blood flow after treatment).

Agree to attend follow-up visits for 2 years.

Patients will be excluded if:

They are pregnant/lactating, have severe vessel calcification that prevents treatment, or have acute limb ischemia/thrombosis.

They have a history of stroke in the past 60 days, contraindications to blood-thinning medications, or a life expectancy of less than 2 years.

How is the study conducted? This is a prospective, multicenter cohort study (observing patients over time) conducted at multiple university-affiliated hospitals in China. A total of 578 eligible patients will be enrolled over approximately 2 years.

Treatment assignment:

Doctors will choose either DCB or DES based on clinical judgment and real-world practice:

DCB group: The narrowed area is first expanded with a standard balloon, then treated with a paclitaxel-coated balloon (to deliver medication to the vessel wall). A bare-metal stent may be used if needed (e.g., if the vessel tears or remains too narrow after DCB treatment).

DES group: After initial balloon expansion, a paclitaxel-eluting stent (a stent that slowly releases medication) is implanted to cover the entire narrowed area.

Follow-up:

Patients will be checked at 1, 3, 6, 12, and 24 months after treatment. Tests will include ultrasound (to check vessel patency), ankle-brachial index (ABI, a measure of blood flow), and assessments of symptoms and adverse events.

What are the study's key goals?

Primary goal (main outcome):

To compare the rate of clinically driven target lesion revascularization (CD-TLR) at 24 months. CD-TLR means needing repeat procedures (e.g., balloon angioplasty or stenting) on the treated area because of worsening symptoms or reduced blood flow.

Secondary goals:

Rates of major adverse limb events (MALE, including major leg amputation).

Vessel patency (whether the treated area stays open):

Primary patency: The vessel remains open without repeat intervention. Secondary patency: The vessel stays open after additional interventions if needed.

Improvement in symptoms and blood flow (measured by ABI and Rutherford class). Stent fracture rate (for DES patients) and safety outcomes (e.g., 30-day death, bleeding, heart attack, or organ function decline).

Is the study safe and regulated? The study has been approved by the Medical Ethics Committee of the Affiliated Hospital of Chengdu University of Traditional Chinese Medicine (Approval No. 2020KL-078) and follows the Declaration of Helsinki (international ethical standards for medical research).

It is registered on ClinicalTrials.gov (NCT04675632) and results will be published in a peer-reviewed medical journal.

Why is this study important? By directly comparing DCBs and DESs-two of the most advanced treatments for femoropopliteal ISR-this study will provide high-quality evidence to help doctors make better treatment decisions. For patients, this means more personalized, effective care that reduces the need for repeat procedures and improves quality of life.

For healthcare providers, the results will clarify which treatment works best for different patients (e.g., those with complex lesions) and optimize endovascular strategies for ISR.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age > 18 years. (2) Willing and able to provide informed consent. (3) Rutherford Clinical Category 2-5. (4) Presence of ≥50% stenosis and/or occlusion (>30 days post-implantation) in a superficial femoral artery stent, located from at least 1cm distal to the origin of the profunda femoris artery to at least 1cm proximal to the femoral intercondylar notch.

  (5) The target lesion must be within the stented segment or extend no more than 3cm proximal or distal to the stent.

  (6) Planned treatment with either a DCB (with provisional BMS stenting) or a DES.

  (7) Total target lesion length ≤30 cm. (8) At least one patent runoff vessel below the knee. (9) Patient is committed to participate in follow-up visits at 1, 3, 6, 12, and 24 months.

Exclusion Criteria:

* (1) Pregnancy or lactation. (2) Rutherford Category 0 or 6. (3) Severe calcification of the target lesion precluding PTA. (4) Acute ischemia and/or acute thrombosis in the target limb. (5) Untreated hemodynamically significant aorto-iliac stenotic disease. (6) Target lesion stenosis <50%. (7) Target lesion length >30 cm. (8) History of cerebrovascular accident within 60 days prior to the procedure. (9) Contraindication to antiplatelet, anticoagulant, or thrombolytic therapy. (10) Inability or unwillingness to provide informed consent. (11) Life expectancy of less than 2 years or other factors making follow-up unlikely.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinically-Driven Target Lesion Revascularization (CD-TLR) | 24 months post-procedure
Clinically-Driven Target Lesion Revascularization (CD-TLR) | 24 months post-procedure
  CD-TLR is defined as any repeat percutaneous or surgical intervention performed on the target lesion (including areas 3 cm proximal and distal to the device edge) due to clinical symptoms and/or a significant drop in functional indices. The primary endpoint assesses the absence of such revascularization in the study population.

IPD SHARING:
Plan to Share IPD: Undecided